CLINICAL TRIAL: NCT06435689
Title: Etude et Modulation de la réponse Immunitaire Dans Les Cancers COlorectaux Primaires et METastatiques
Brief Title: Study and Modulation of Immune Responses in Primary and Metastatic Colon Cancers
Acronym: I-COMET
Status: Not yet recruiting | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: APHP231721
Record Dates: First submitted 2024-05-26; First posted 2024-05-30 (Actual); Last update posted 2024-05-30 (Actual); Status verified 2024-05

CONDITIONS: Colon Cancer; Peritoneal Carcinoma
Keywords: Organoids; T-cells; Metastasis; Immunotherapies
MeSH Terms: conditions — Colonic Neoplasms; Neoplasm Metastasis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood and surgical specimen sampling the day of surgery (primary tumor and metastases if applicable)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients undergoing surgery for the treatment of primary and/or metastatic colorectal cancers
  Interventions: Other: Sampling

INTERVENTIONS:
Other: Sampling — Blood and surgical specimen sampling the day of surgery

SUMMARY:
Colorectal cancer (CRC) is the 3rd most common cancer in France. Treatment of CRC relies primarily on surgical removal of the primary tumor and chemotherapy is the current standard of care for synchronous metastatic disease. Overall survival remains strongly correlated with the tumor stage at the time of surgery, from 90% at five years for localized disease (stages 1 and 2), to around 20% for metastatic forms of the disease (stage 4). Recent research in cancer highlights the role of the immune system in the development, evolution and fate of tumors. Understanding the nature of interactions between different immune cells infiltrating the tumor is important for the development of innovative therapies. Recently, the consensus molecular classification of CRC confirmed the importance of the immune response in CRC by showing that a "high immune response" is a good prognostic indicator for patients with this pathology. However, immunotherapies are effective for only a minority of patients with metastatic CRC. Indeed, anti Programmed cell Death 1 (anti-PD-1), -PD-L1 immune checkpoint blocking antibodies have only shown effectiveness in patients with microsatellite instability (MSI), which only represents 5% of metastatic CRCs.

Thus, the aim of this study is to better understand the role of the immune system on the development of CRC and its possible modulation to treat or prevent metastatic recurrences.

ELIGIBILITY:
Inclusion Criteria:

* Male or female 18 years of age or older
* Diagnosis of colorectal adenocarcinoma
* Scheduled resection of tumor and/or metastasis(es)

Exclusion Criteria:

* Patient's opposition to research
* Patients under guardianship
* The following situations

  1. Persons unable to understand and/or read the information leaflet
  2. Patient with one of the following functions: Investigator or co-investigator, research assistant, pharmacist, study coordinator or, having any involvement in the study
  3. Non-cooperative or potentially non-compliant person for the study and its procedures with foreseeable difficulties in regular follow-up over 5 years.
  4. Non-affiliation with a social security scheme, Couverture Médicale Universelle or any equivalent scheme.
* Pregnant or breast-feeding women.
* HIV-positive patients.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing surgery for the treatment of primary and/or metastatic colorectal cancers
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2024-06-15 (Estimated); Primary Completion 2025-06-15 (Estimated); Study Completion 2039-06-15 (Estimated)

PRIMARY OUTCOMES:
Effectiveness of immunotherapies in a co-culture model | At 1 year
  Characterize effective immunotherapies in colorectal cancers by demonstrating their effectiveness in a co-culture model between cancer cells and autologous T cells.

SECONDARY OUTCOMES:
Evaluation of transcriptomic differences | At 5 years
  Evaluation of transcriptomic differences between tissues or cells from the healthy mucosa compared to those from the primary or metastatic tumor: sequencing of mRNA in the two types of mucosa and comparison of mRNA expression profiles between the latter.
Evaluation of proteomic differences | At 5 years
  Evaluation of proteomic differences between tissues or cells from the healthy mucosa in comparison to those from the primary tumor by:
  multiplexed immunodetection in situ in tissues detection and dosage of proteins in culture supernatants (ELISA), in a co-culture model between cancer cells and autologous T cells, with or without modulation of a pathway targeting the T lymphocyte response by immunotherapy.
Evaluation of the T Cell Receptor (TCR) repertoire | At 5 years
  Evaluation of the TCR repertoire by sequencing, carried out from:
  patient blood, DNA from cancerous tissues and healthy mucosa DNA from the co-culture between cancer cells and autologous T cells, with or without modulation of a pathway targeting the T lymphocyte response by immunotherapy

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - Hôpital Saint Louis - gastoenterology, Paris
  - Hôpital Saint Louis - visceral, oncological and endocrine surgery, Paris